CLINICAL TRIAL: NCT05802173
Title: A Randomized, Double-blind, Vehicle-controlled, Parallel Group, Multi-dose Study to Evaluate the Efficacy and Safety of TDM-105795 in Male Subjects With Androgenetic Alopecia
Brief Title: Study of TDM-105795 Following Topical Administration in Male Subjects With Androgenetic Alopecia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Technoderma Medicines Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 239-11651-203
Record Dates: First submitted 2023-03-14; First posted 2023-04-06 (Actual); Results first posted 2025-11-12 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2024-11

CONDITIONS: Alopecia, Androgenetic
MeSH Terms: conditions — Alopecia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TDM-105795 topical solution, 0.0025% (Experimental): Daily dose of 0.0025% of TDM-105795 topical solution
  Interventions: Drug: TDM-105795, 0.0025%
- TDM-105795 topical solution, 0.02% (Experimental): Daily dose of 0.02% of TDM-105795 topical solution
  Interventions: Drug: TDM-105795, 0.02%
- TDM-105795 topical vehicle solution (Placebo Comparator): Daily dose of placebo for TDM-105795 topical solution
  Interventions: Drug: TDM-105795 topical vehicle solution

INTERVENTIONS:
Drug: TDM-105795, 0.0025% — The assigned drug will be applied once daily for 16 weeks, with application to the scalp focusing on the regions that are bald and thinning.
  Arms: TDM-105795 topical solution, 0.0025%
Drug: TDM-105795, 0.02% — The assigned drug will be applied once daily for 16 weeks, with application to the scalp focusing on the regions that are bald and thinning.
  Arms: TDM-105795 topical solution, 0.02%
Drug: TDM-105795 topical vehicle solution — The assigned placebo will be applied once daily for 16 weeks, with application to the scalp focusing on the regions that are bald and thinning.
  Arms: TDM-105795 topical vehicle solution

SUMMARY:
Randomized, double-blind, vehicle-controlled, parallel group, multi-dose study of TDM-105795 in male subjects with androgenetic alopecia

DETAILED DESCRIPTION:
Protocol 239-11651-203 is a Phase 2 study entitled "A Randomized, Double-Blind, Vehicle-Controlled, Parallel Group, Multi-Dose Study to Evaluate the Efficacy and Safety of TDM-105795 in Male Subjects with Androgenetic Alopecia" Eligible subjects will be randomized (1:1:1) to 1 of the 3 groups (low dose vs high dose vs placebo) and treated for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

To enter the study, a subject must meet the following criteria:

1. Subject is male, 18-55 years old.
2. Subject has provided written informed consent.
3. Subject has a clinical diagnosis of mild to moderate androgenetic alopecia (AGA) in temple and vertex region with a score of IIIv, IV, or V on the Modified Norwood-Hamilton Scale.
4. Subject, in the investigator's opinion, is in good general health and free of any disease state or physical condition that might impair evaluation of AGA or exposes the subject to an unacceptable risk by study participation.
5. Subject has normal renal, thyroid, and hepatic function as determined by the Visit 1/Screening laboratory results in the opinion of the investigator.
6. Subject is a non-smoker, defined as not having smoked or used any form of tobacco or non-tobacco products containing nicotine in more than 4 months before Visit 2/Baseline.
7. Subject is willing to maintain the same hair style, hair length, and hair color throughout the study.
8. Subject agrees to continue his other general hair care products and regimen for at least 2 weeks prior to Visit 2/Baseline, and through the entire study.
9. Subject is willing and able to apply the investigational product (IP) as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
10. Subjects who are sexually active with a female partner and are not surgically sterile ( vasectomy performed at least 6 months prior to treatment) must agree to refrain from sperm donation for at least 90 days after administration of their last dose of IP and inform their non-pregnant female sexual partner to use a highly effective form of birth control1 as described in the informed consent form. Note: Female partner must be confirmed according to subject to be non-pregnant at Visit 1/Screening and Visit 2/Baseline or at the visit when a subject identifies a new sexual partner.

Exclusion Criteria:

A subject is ineligible to enter the study if he meets 1 or more of the following criteria:

1. Subject has any dermatological disorders of the scalp on the regions that are bald and thinning with the possibility of interfering with the application of the IP or examination method, such as fungal or bacterial infections, seborrheic dermatitis, psoriasis, eczema, folliculitis, scars, or scalp atrophy.
2. Subject has history or active hair loss due to diffuse telogen effluvium, alopecia areata, scarring alopecia, trichotillomania, or conditions/diseases other than AGA.
3. Subject has any skin pathology or condition (e.g., uncontrolled thyroid disease, certain genetic disorders that involve hair growth or patterns) that, in the investigator's opinion, could interfere with the evaluation of the IP or requires use of interfering topical, systemic, or surgical therapy.
4. Subject has any visible inflammatory skin disease, injury, or condition of their scalp that could compromise subject safety and/or interfere with the evaluation of local or systemic assessments performed during the study.
5. Subject has history (within 6 months of Visit 1/Screening) of severe dietary or weight changes or history of eating disorder(s), which has resulted in hair loss, in the opinion of the investigator.
6. Subject has a history of scalp reduction or notable trauma with related scarring, hair transplants, and/or hair weaves.
7. Subject has a known or suspected malignancy excluding cutaneous basal cell carcinoma or cutaneous squamous cell carcinoma not located within the treatment area.
8. Subject has a positive blood screen for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg), or hepatitis C antibody.
9. Subject has any condition, which, in the investigator's opinion, would make it unsafe for the subject to participate in this study, including clinically significant abnormal laboratory, or 12-lead electrocardiogram (ECG) findings during the screening period or Visit 2/Baseline prior to dosing of the IP.
10. Subject has used any topical scalp treatments for hair growth including minoxidil, hormone therapy, anti-androgen, or other agents known to affect hair growth within 12 weeks of Visit 2/Baseline.
11. Subject has used any topical scalp over-the-counter (OTC) or cosmetic treatments known or reasonably believed to affect hair growth (e.g., brands such as Aminexil, Maxilene, Nioxin, Foltene) or hair growth products with saw palmetto, copper, etc. within 4 weeks of Visit 2/Baseline.
12. Subject has used any topical scalp treatments that may have ancillary effects on hair growth including, but not limited to, corticosteroids, pimecrolimus, tacrolimus, and retinoids within 4 weeks of Visit 2/Baseline.
13. Subject has had any scalp procedures, including surgical, laser, light or energy treatments, micro-needling, etc. within 6 months of Visit 2/Baseline.
14. Subject has had platelet rich plasma (PRP) procedures on the scalp at any time.
15. Subject has used systemic beta blockers, cimetidine, ketoconazole, diazoxide, or corticosteroids (including intramuscular and intralesional injections) within 12 weeks of Visit 2/Baseline. Inhaled, intranasal, or ocular corticosteroids are allowed if use is stable. Stable is defined as doses and frequency unchanged for at least 4 weeks prior to Visit 2/Baseline.
16. Subject has used systemic retinoids, isotretinoin, vitamin A intake above 10,000 IU per day, or cyclosporine therapy within 6 months of Visit 2/Baseline.
17. Subject has used finasteride (e.g., Propecia®), dutasteride, minoxidil (oral), or similar products within 6 months of Visit 2/Baseline.
18. Subject has used chemotherapy or cytotoxic agents within 12 months of Visit 2/Baseline.
19. Subject has had radiation of the scalp at any point.
20. Subject has used any other systemic therapy, which in the opinion of the investigator, may materially affect the subject's hair growth, including, but not limited to, vitamin or homeopathy supplement hair growth or hair health products or other steroid hormones (in any form), including anabolic steroids.
21. Subject is currently enrolled in an investigational drug, biologic, or device study.
22. Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days or 5 half-lives, whichever is longer, prior to Visit 2/Baseline.
23. Subject has previously been treated with the IP.
24. Subject has a history of prescription drug abuse, or illicit drug use within 6 months prior to Visit 1/Screening.
25. Subject has a history of alcohol abuse according to medical history within 6 months prior to Visit 1/Screening.
26. Subject has a positive screen for alcohol or drugs of abuse at Visit 1/Screening or Visit 2/Baseline.
27. Subject has signs or symptoms consistent with Coronavirus Disease-19 (COVID-19) at Visit 1/Screening or Visit 2/Baseline or has been diagnosed with COVID-19 within 4 weeks of Visit 1/Screening.
28. Subject has a history of sensitivity to any of the ingredients in the IP or tattoo ink.
29. Subject is known to be noncompliant or is unlikely to comply with the requirements of t the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 71 (Actual)
Dates: Start 2023-03-06 (Actual); Primary Completion 2023-11-08 (Actual); Study Completion 2024-01-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J. Piacquadio, M.D., Study Director — Therapeutics Incorporated
Locations (13):
- United States (13):
  - Site 12, North Little Rock, Arkansas
  - Site 4, Rolling Meadows, Illinois
  - Site 7, Plainfield, Indiana
  - Site 11, Baton Rouge, Louisiana
  - Site 13, New Orleans, Louisiana
  - Site 10, Minneapolis, Minnesota
  - Site 9, New Brighton, Minnesota
  - Site 3, Portland, Oregon
  - Site 5, Knoxville, Tennessee
  - Site 8, Murfreesboro, Tennessee
  - Site 1, Austin, Texas
  - Site 6, College Station, Texas
  - Site 2, Norfolk, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 71 participants randomized in the study and were evaluable for safety analyses.
Period: Overall Study
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Started | 26 | 23 | 22
Completed | 23 | 16 | 18
Not Completed | 3 | 7 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 6 | 4
Not completed — non-compliance | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution | Total
Number analyzed (Participants) | 26 | 23 | 22 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (8.84) | 40.7 (9.73) | 40.8 (9.38) | 40.9 (9.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 26 | 23 | 22 | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3 | 6
  Not Hispanic or Latino | 23 | 23 | 19 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 5 | 5 | 11
  White | 24 | 15 | 15 | 54
  More than one race | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Non-vellus Target Area Hair Count (TAHC)
Description: Collection of non-vellus target area hair count results at week 16
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: hair count
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 26 | 23 | 22
hair count | 20.3 (29.40) | 22.4 (18.59) | 14.0 (17.59)

2. Primary Outcome: Evaluation of Treatment Benefit
Description: Collection of hair growth assessment (HGA) questionnaire at week 16. Scalp hair growth will be compared from Baseline using the following 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 26 | 23 | 22
Participants
  Slightly to moderately decreased | 4 | 3 | 1
  No change | 10 | 5 | 9
  Slightly to moderately increased | 9 | 8 | 8
  Missing | 3 | 7 | 4

3. Secondary Outcome: Change in Non-vellus Target Area Hair Width (TAHW)
Description: Collection of non-vellus target area hair width results at week 16
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 21 | 13 | 15
microns | -1.27 (2.30) | -2.18 (2.00) | -1.27 (2.20)

4. Secondary Outcome: Change in Non-vellus Target Area Hair Darkness (TAHD)
Description: Non-vellus Target Area Hair Darkness (TAHD) results at week 16. Scale is a gray scale, 0(white) to 255(black) measured in a 1 cm2 area. Positive mean change is a better outcome.
Time Frame: 16 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 21 | 13 | 15
score on a scale | 4.6 (12.27) | 3.2 (15.52) | -3.6 (14.33)

5. Secondary Outcome: Hair Growth Index (HGI) Questionnaire
Description: Subject's evaluation of treatment benefit via the hair growth index (HGI) questionnaire at week 16. Scalp hair growth will be compared from Baseline using the following 7-point scale: much less (-3), moderately less (-2), slightly less (-1), the same amount (0), slightly more (1), moderately more (2), and much more (3).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 26 | 23 | 22
Participants
  Slightly to moderately less scalp | 8 | 6 | 7
  Same amount | 10 | 4 | 8
  Slightly to moderately more scalp | 5 | 6 | 3
  Missing | 3 | 7 | 4

6. Secondary Outcome: Evaluation of Investigator's Global Assessment (IGA) Grade
Description: Collection of IGA grade at week 16. The Canfield Review application will be used. The evaluator will assess the subject's scalp hair growth using the following 7-point scale: greatly decreased (-3), moderately decreased (-2), slightly decreased (-1), no change (0), slightly increased (1), moderately increased (2), and greatly increased (3).
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 26 | 23 | 22
Participants
  slightly to moderately decreased | 1 | 3 | 0
  No change | 9 | 5 | 12
  slightly to moderately increased | 13 | 8 | 6
  Missing | 3 | 7 | 4

7. Other Pre Specified Outcome: Number of Participants With Any Local and Systemic Adverse Events (AEs)
Description: Collection of adverse events
Time Frame: 20 weeks
Measure: Number; unit: participants
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 26 | 23 | 22
participants
  Subjects with any TEAE | 8 | 6 | 7
  Subjects with any treatment related TEAE | 1 | 5 | 1
  Subjects with any serious TEAE | 0 | 0 | 0

8. Other Pre Specified Outcome: Number of Subjects With Presence (and Severity) of Local Skin Reactions (LSRs)
Description: Collection of local skin reactions at day 1, week 2, week 4, week 8, week 12, and week 16
Time Frame: 16 weeks
Measure: Number; unit: participants
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
Number analyzed (Participants) | 26 | 23 | 22
participants
  Erythema | 10 | 10 | 2
  Edema | 3 | 1 | 2
  Erosion | 1 | 1 | 0
  Scaling | 1 | 4 | 0
  Pruritus | 1 | 5 | 2
  Burning/Stingling | 3 | 3 | 0

ADVERSE EVENTS:
Time Frame: 16 weeks
Arm/Group | TDM-105795 Topical Solution, 0.0025% | TDM-105795 Topical Solution, 0.02% | TDM-105795 Topical Vehicle Solution
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/23 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/23 | 0/22
Other Adverse Events (participants affected / at risk) | 8/26 | 6/23 | 7/22
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TDM-105795 Topical Solution, 0.0025% (N=26) | TDM-105795 Topical Solution, 0.02% (N=23) | TDM-105795 Topical Vehicle Solution (N=22)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 1
Application site erythema (General disorders) | 0 | 1 | 0
Application site irritation (General disorders) | 1 | 0 | 0
Application site pain (General disorders) | 0 | 1 | 0
Application site pruritus (General disorders) | 1 | 2 | 0
Fatigue (General disorders) | 0 | 1 | 0
Application site folliculitis (Infections and infestations) | 0 | 2 | 0
COVID-19 (Infections and infestations) | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Scratch (Injury, poisoning and procedural complications) | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Synovial cyst (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 1 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator and all employees and coworkers involved with this study shall not disclose or use for any purpose other than performance of the study, any data, records, or other unpublished, confidential information disclosed to those individuals for the purpose of the study. Prior written agreement from TI or the Sponsor must be obtained for the disclosure of any said confidential information to other parties.

DOCUMENTS (2):
  • Study Protocol (2022-11-30): https://cdn.clinicaltrials.gov/large-docs/73/NCT05802173/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-13): https://cdn.clinicaltrials.gov/large-docs/73/NCT05802173/SAP_001.pdf